CLINICAL TRIAL: NCT00348192
Title: A Double-Blind, Randomised, Placebo-Controlled, Parallel Group Study to Investigate the Effects of SB-742457, Donepezil and Placebo on Cognition in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: SB-742457 And Donepezil In Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZ3106242
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; cognition global functioning; symptomatic; SB-742457
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-benzenesulfonyl-8-piperazin-1-ylquinoline; Donepezil

INTERVENTIONS:
Drug: SB-742457
Drug: donepezil
  Other Names: SB-742457

SUMMARY:
The purpose of this study is to find out if SB-742457 is a safe treatment and what effects it has on the symptoms of mild to moderate Alzheimer's Disease. SB-742457 is a new treatment which is thought to increase the levels of certain chemicals in the brain that are often decreased in patients with Alzheimer's Disease.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of probable mild-to-moderate Alzheimer's Disease as determined by the NINCDS-ADRDA and DSM-IV criteria with an MMSE score of 12-24.
* Subjects and their caregivers must provide informed consent prior to study entry.
* Adequate blood pressure and laboratory values.

Exclusion criteria:

* Females of child-bearing potential.
* Have other causes of dementia such as vascular damage, depression, bipolar affective disorder, schizophrenia, syphilis, vitamin B12 deficiency or thyroid deficiency.
* Subjects taking medication for Alzheimers disease or centrally acting agents which might impact study outcomes.
* Subjects taking agents for which there is a theoretical risk of interaction with SB-742457 or donepezil.
* Subjects with conditions which might be exacerbated by exposure to donepezil.
* Subjects with known hypersensitivity to sunlight or seizures.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-05

PRIMARY OUTCOMES:
Change in cognition and function after 24 weeks.

SECONDARY OUTCOMES:
Change in behavioral symptoms, activities of daily living and caregiver burden after 24 weeks Changes in all symptoms at 8 and 12 weeks Safety and tolerability PK (pharmacokinetic) profiling. Efficacy related to ApoE and HTR6 status

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (20):
- Austria (2):
  - GSK Investigational Site, Hall in Tirol
  - GSK Investigational Site, Vienna
- Bulgaria (2):
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Chile (3):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Providencia / Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (5):
  - GSK Investigational Site, Ostfildern, Baden-Wurttemberg
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Baesweiler, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- GSK Investigational Site, Bratislava, Slovakia
- United Kingdom (3):
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Swindon
  - GSK Investigational Site, West of Scotland Science Park, Glasgow

REFERENCES:
- [Derived] Maher-Edwards G, Dixon R, Hunter J, Gold M, Hopton G, Jacobs G, Hunter J, Williams P. SB-742457 and donepezil in Alzheimer disease: a randomized, placebo-controlled study. Int J Geriatr Psychiatry. 2011 May;26(5):536-44. doi: 10.1002/gps.2562. Epub 2010 Sep 24. PMID 20872778